CLINICAL TRIAL: NCT04234022
Title: Zn-DDC to Target Hypoxia-NFkappaB-CSCs Pathway and Improve the Treatment Outcomes of Haematological Malignancies - A Translation Bench Study
Brief Title: Zn-DDC to Target Hypoxia-NFkappaB-CSCs Pathway in Multiple Myeloma
Status: Recruiting | Type: Observational
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Collaborators: University of Wolverhampton (Other)
Responsible Party: Sponsor
Other Study IDs: 2019HAE109
Record Dates: First submitted 2020-01-15; First posted 2020-01-21 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Zn-DDC: samples to be exposed with Zn-DDC (Imuthiol) alone
  Interventions: Drug: Zn-DDC
- Lenalidomide with Zn-DDC: samples to be exposed with Lenalidomide in combination with Zn-DDC
  Interventions: Drug: Lanalidomide with Zn-DDC
- Pomalidomide with Zn-DDC: samples to be exposed with Pomalidomide in combination with Zn-DDC
  Interventions: Drug: Pomalidomide with Zn-DDC

INTERVENTIONS:
Drug: Zn-DDC — Zn-DDC added to myeloma samples for culturing
  Groups: Zn-DDC
Drug: Lanalidomide with Zn-DDC — Lanalidomide with Zn-DDC added to myeloma samples for culturing
  Groups: Lenalidomide with Zn-DDC
Drug: Pomalidomide with Zn-DDC — Lanalidomide with Zn-DDC added to myeloma samples for culturing
  Groups: Pomalidomide with Zn-DDC

SUMMARY:
The outlook for patients with haematological malignancies remains challenging. It has been shown in some early cancer studies that a particular drug called Zn-DDC otherwise known as Imuthiol is highly toxic to cancer stem cells. Imuthiol has been intravenously used in clinical trials with an excellent safety record. Recent novel therapy and immunotherapy in haematological malignancies have improved outcome and survival but come with an increasing cost burden. Imuthiol could be an ideal affordable drug to study on it's own as well as in combination with other drugs in myeloma and other haematological malignancies. This may lead to potential combination therapies which will be very effective as well as affordable in the future. There is the need to look to see if this drug, Imuthiol and along with complementary drugs lenalidomide (Revlimid) and pomalidomide (Pomalyst) can help in haematological malignancy treatment. In order to do this there is the need to see how the cancer cells respond to the drugs in the laboratory before being able to trial the drug (or combination of drugs) out for treatment. The success of this study may lead to quick translation of Imuthiol into haematological malignancy treatment.

DETAILED DESCRIPTION:
Up to 60 myeloma bone marrow samples from Myeloma patients and 10 bone marrow samples from other haematological malignancy samples (Acute leukaemia's) at Diagnosis and Relapse will be tested.

Patients attending haematology clinics at New Cross Hospital will be reviewed for eligibility of the study by the clinician and if they meet the recruitment criteria, they will be approached to participate at clinic.

After informed consent, participants will be asked to donate an additional 2-3ml sample of bone marrow in a single aliquot for the purpose of this study whilst undergoing a bone marrow aspirate as part of their routine clinical care at diagnosis and relapse.The single aliquot will be sent to the University of Wolverhampton for analysis.

Specific clincial data will be collected at the time of diagnosis and relapse:

* Diagnosis
* Date diagnosed
* Disease stage
* Relapse status
* Age
* Sex
* Previous treatments
* Date of marrow sample
* Marrow trephine
* Marrow liquid The clinical data set will remain at The Royal Wolverhampton NHS Trust whilst analysis of the samples takes place. Once the samples have been analysed, the clinical data will then be released to determine relapsed or refractory disease and correlation with the in vitro data.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with haematological malignancy - either myeloma or acute leukaemia
* Patients must be 18 years or over
* Patients must be willing and able to give informed consent

Exclusion Criteria:

* Pregnant patients will not be entered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 60 myeloma bone marrow samples from Myeloma patients and 10 bone marrow samples from other haematological malignancy samples (Acute leukaemia's) at Diagnosis and Relapse will be tested.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Imuthiol and zinc efficacy | 7 days
  examine the cyctotoxicity of Imuthiol and zinc in combination with other drugs
Cell kill and determination of IC50 (inhibitory concentration) and apoptotic pathways involved | 7 days
  Cell kill and determination of IC50 (inhibitory concentration) and apoptotic pathways involved

CONTACTS AND LOCATIONS:
Overall Officials: Supratik Basu, Principal Investigator — The Royal Wolverhampton NHS Trust
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No